CLINICAL TRIAL: NCT02270086
Title: Evaluating Bacterial Response Throughout Sarcoma Management Using An Optically Tracked, Hand-Held Fluorescent Imaging Device
Brief Title: Evaluating Bacterial Response in Sarcoma Management Using Fluorescence Imaging
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1038
Record Dates: First submitted 2013-11-18; First posted 2014-10-21 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Soft Tissue Sarcoma; Wounds
MeSH Terms: conditions — Sarcoma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sarcoma patient: Patient diagnosed with soft tissue sarcoma and receiving preoperative radiotherapy.

SUMMARY:
The investigators have recently developed an innovative optical molecular imaging platform (called PRODIGI) based on high-resolution fluorescence and white-light technologies in a hand-held, real-time, high-resolution, non-invasive format. PRODIGI offers a non-contact means of obtaining instantaneous image-based measurements of diagnostically-relevant biological and molecular information of a wound and surrounding skin tissues for the first time and could have significant impact on improving conventional wound care, management, and guidance of intervention. In preliminary preclinical testing, the investigators have discovered that when wounds are illuminated by violet/blue light, endogenous collagen in the connective tissue matrix emit a characteristic green fluorescent signal, while most pathogenic bacterial species emit a unique red fluorescence signal due to the production of endogenous porphyrins. Therefore, with autofluorescence imaging, no exogenous contrast agents are needed during imaging, making this approach particularly appealing as a diagnostic imaging method for clinical use.

In the context of this study, PRODIGI is used to assess wound complications in patients diagnosed with soft tissue sarcoma and treated with pre-operative radiotherapy. Both pre- and postoperative external beam radiotherapy combined with limb salvage surgery have similarly high rates of local control in the management of extremity soft tissue sarcoma. The main acute side effect associated with preoperative radiotherapy is wound healing complications. Wound care overall is a major clinical challenge and presents an enormous burden to health care worldwide. The objective of this clinical study is to determine if PRODIGI coupled with an optical tracking platform has clinical utility in identifying, quantitatively measuring and longitudinally tracking bacterial imbalance on the patient's intact skin surface at the location of the surgical resection site for adult patients with lower limb soft tissue sarcoma treated with preoperative intensity-modulated radiation therapy and limb salvage surgery and, further, to investigate whether this bacterial imbalance is related to radiotherapy dose and wound complications.

DETAILED DESCRIPTION:
Optical Tracking System

For this study, PRODIGI was combined with a commercial optical tracking system (OTS, Polaris, NDI Medical, Waterloo, Ontario, Canada) to track the movement of the device in space relative to a patient over time. This addition is in the form of an infrared-light camera, which tracks four IR reflective spheres (NDI Medical, Waterloo, Ontario, Canada) that are fixed to the external housing of PRODIGI device.

The OTS has been described previously. Briefly, it consists of optical tracking technology, which provides 6 degrees of freedom (x, y, z, pitch. yaw, roll), attached to the camera along with software developed in house to register and visualize the tracked camera pose relative to a previously acquired radiological volumetric image data. The in-house software platform GTxEyes performs tracking and navigation of the imaging camera, camera calibration (including any image distortion), registration of the camera coordinates with respect to the CT images, and co-visualization (e.g. visual overlay) of the camera and CT images. Radiation dose planning information can also be spatially co-registered and overlaid with the hybrid optical-CT images/videos using methods described previously by our group.

After loading a CT image of the patient, the OTS is registered to the CT coordinate space by identification of known fiducials using a conventional pointer tool. With registration complete, the coordinates of the PRODIGI camera can be tracked in real time relative to the CT image. Viewing options include orthogonal views through the CT image, corrected PRODIGI image and a virtual image based on the CT surface rendering viewed from the perspective of a virtual camera at the PRODIGI coordinates. Radiation dose can be displayed on the real and virtual camera views as either isodose lines or colorwash.

Patient Population

Patients will be recruited from the Princess Margaret Cancer Centre, University Health Network (Ontario, Canada) sarcoma clinic to be treated with pre-operative external beam RT followed by surgical resection of lower limb soft-tissue sarcoma. Informed consent was obtained according to institutional Research Ethics Board (REB) requirements and Good Clinical Practice (GCP) (ClinicalTrials.gov NCT02270086). Patients with pre-existing skin issues, who received prior radiotherapy or required chemotherapy were not eligible to the study.

Imaging Procedures

At the radiotherapy planning stage, a CT scan of the patient sarcoma site is acquired for standard treatment planning purposes. Prior to the CT scan, small radio-opaque fiduciary markers (Suremark TM skin marking labels) were placed on the patient's six radiation treatment setup points, making the <1 mm diameter points easy to identify in the CT images. After the CT scan, these markers were replaced with ink tattoos and used during radiation treatment to align the patient with radiation therapy machine reference frame. In addition to the CT fiducial markers placed at the treatment setup points, a flexible radio-opaque wire was overlaid on the planned surgical incision. This enabled localization of the entire surgical scar during the radiation treatment plan procedure. A radiotherapy stereotactic mask was also made at that stage. Following CT simulation scan acquisition, an appropriate radiotherapy plan was designed as per institutional clinical standard guidelines.

Imaging with PRODIGI and the OTS was performed throughout the sarcoma management, i.e. during radiotherapy and in the operating room. Imaging was performed at three time points during RT: fractions 0, 12 and 25, i.e. at the beginning, middle and end of the treatment. Four out of six treatment setup points marked with radio-opaque fiduciary markers on the CT scans were used to perform the optical to CT co-registration. An optically-tracked pointer tool using four IR reflective spheres (identical to the ones fixed to the PRODIGI system) was used to register the patient in space with respect to the IR camera. For this, the pointer was placed sequentially on each tattoo mark, identified and spatially registered by the tracking IR camera and visualized in real-time on the CT scans using the custom-built software GTxEyes. The locations of the tattoo points in the optical tracking coordinate system were then registered to the corresponding points in the CT image using the fiduciary CT markers. Once registration was completed, the planned surgical scar was drawn on the patient's skin with a marker by superimposing the optically-tracked pointer on the scar visible on the CT scans. An imaging session consisted of both WL and corresponding AF imaging of the planned skin surgical incision and surrounding tissue. Room lights were turned off during AF imaging to avoid background signal and artifacts. The four reflective spheres on the PRODIGI device were pointed towards the IR camera to ensure proper tracking in 3D during the entire session.

To perform PRODIGI imaging in the operating room, a sterilization method approved by UHN's control and processing department using a sterile drape was found to be the most effective way to ensure proper sterile conditions without damaging the instrument or affecting its performance. An elongated sterile drape (Cardinal Health Canada, 29-59029) was used to cover the entire PRODIGI imaging system, i.e. the camera and electrical power cord. Six strong neodymium magnets (Super Magnets, 8 mm diameter) were embedded into the emission filter slider and six corresponding magnets were autoclaved prior to each use and placed on the outside of the drape to hold it in place to avoid image quality degradation. Steri-strips (3M, R1547) were applied on the outside of the draped device to tighten the drape around the IR reflective spheres to insure adequate tracking during imaging. Imaging was performed at five time points: before and after sterilization of the surgical site (OR1, OR2), once the flap was raised (OR3), after tumor excision (OR4) and after closure (OR5).

The combined WL and AF images were part of a superset of data recorded using the tracking system. The superset also included preoperative patient CT and the patient's RT dose volume. A skin surface model was generated from the patient's CT, where each surface point held a quantitative tuple that contained the surface normal vector, the RT dose, the WL scalar, the AF scalar, and the camera pose corresponding to the AF scalar. Overlay of WL and AF images on the skin surface model was visualized using the software ParaView.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven soft tissue sarcoma following review by local reference pathologist.
* Deemed appropriate for preoperative radiotherapy and limb salvage surgery following patient assessment by a radiation oncologist and surgical oncologist and after discussion between both specialists.
* Lesion lies distal to the iliac crest and proximal to the ankle.
* Lesion is primary or locally recurrent. Patient may have undergone excisional biopsy with positive margins at a referring hospital and are eligible following discussion among the surgical oncologists and radiation oncologists that IMRT is an acceptable treatment for that case.
* Patient is aged 18 years or older.
* Patient must be available for treatment and follow-up at Mount Sinai Hospital/Princess Margaret Hospital.
* Protocol treatment is to begin within 4 weeks of entry.
* Patients must be capable of giving informed consent, and informed consent must be obtained according to local Research Ethics Board (REB) requirements.

Exclusion Criteria:

* Benign histology.
* Histology generally treated with adjuvant chemotherapy, such as rhabdomyosarcoma, primitive neurectodermal tumor (PNET), soft tissue Ewing's sarcoma or soft tissue osteosarcoma.
* Prior or concurrent malignancy, with the exception of adequately treated basal cell carcinoma of the skin or carcinoma in-situ of the cervix.
* Limb conservation is not appropriate.
* Prior radiotherapy to the local site or chemotherapy.
* Pathological review of total specimen required before the need for irradiation can be assessed.
* Chemotherapy is required as an adjuvant treatment.
* Presence of regional nodal disease or unequivocal distant metastases.
* Other major medical illness deemed to preclude safe administration of protocol treatment or required follow-up.
* Treatment with an investigational drug within 1 month before study enrolment.
* Any contra-indication to routine wound care and/or monitoring.
* Patients with pre-existing skin issues (e.g. melanomas, psoriasis) in areas close to the potential wound(s) that will be studied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted at the Princess Margaret Cancer Centre in Toronto. Patients present with soft tissue sarcoma and receive pre-operative radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of bacterial presence changes by microbiology swabbing tests | Each study visit over the course of 20-25 weeks, i.e. 7-10 study visits
  Microbiology swabbing will be performed during radiotherapy treatments (3 visits), surgery (1 visit) and follow-up appointments (3-6 visits depending on wound healing) to monitor changes in bacterial presence

SECONDARY OUTCOMES:
Complication requiring wound care or second surgery | 6-8 weeks after surgery
  Wound complication is identified 6-8 weeks after surgery, i.e. normal time frame for complete closure of surgical incision

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DaCosta, PhD, Principal Investigator — University Health Network, Toronto; Peter Ferguson, MD, Principal Investigator — University Health Network, Mount Sinai Hospital
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented in a peer-reviewed journal at completion of study